CLINICAL TRIAL: NCT00566644
Title: Prevention of Endometrial Tumors (POET)
Brief Title: Intrauterine Levonorgestrel and Observation or Observation Alone in Preventing Atypical Endometrial Hyperplasia and Endometrial Cancer in Women With Hereditary Non-Polyposis Colorectal Cancer or Lynch Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn due to poor accrual
Sponsor: St George's, University of London (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: CRUK-POET; CDR0000575423 (Registry Identifier: PDQ (Physician Data Query)); EudraCT 2006-001815-30; EU-20784
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-10

CONDITIONS: Endometrial Cancer; Hereditary Non-polyposis Colon Cancer (hmsh2, hmlh1, hpms1, hpms2)
Keywords: endometrial cancer; hereditary non-polyposis colon cancer (hMSH2, hMLH1, hPMS1, hPMS2)
MeSH Terms: conditions — Endometrial Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Observation

INTERVENTIONS:
Device: levonorgestrel-releasing intrauterine system
Other: questionnaire administration
Procedure: observation

SUMMARY:
RATIONALE: The use of intrauterine levonorgestrel may prevent atypical endometrial hyperplasia and endometrial cancer in women with hereditary non-polyposis colorectal cancer or Lynch syndrome. It is not yet known whether intrauterine levonorgestrel and observation are more effective than observation alone in preventing atypical endometrial hyperplasia and endometrial cancer in women with hereditary non-polyposis colorectal cancer or Lynch syndrome.

PURPOSE: This randomized phase III trial is studying intrauterine levonorgestrel and observation to see how well they work compared with observation alone in preventing atypical endometrial hyperplasia and endometrial cancer in women with hereditary non-polyposis colorectal cancer or Lynch syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if treatment with intrauterine levonorgestrel (using the Mirena® intrauterine system [IUS]) reduces the incidence of atypical endometrial hyperplasia (AEH) and endometrial cancer in women with hereditary non-polyposis colorectal cancer or Lynch syndrome.

Secondary

* Determine the age-related incidence of AEH and endometrial cancer in these patients.
* Determine the sensitivity and specificity of transvaginal sonography and endometrial biopsy in detecting AEH and endometrial cancer.
* Determine the premalignant pathway to carcinoma.
* Determine if the Mirena® IUS reduces the rate of therapeutic hysterectomy for AEH or endometrial cancer.
* Determine the psychological benefits or adverse effects from the use of the Mirena® IUS.
* Determine the satisfaction and compliance with screening.
* Determine the extent of adverse effects of the Mirena® IUS and observation.
* Determine the molecular changes associated with pre-malignant changes in the endometrium of these patients, and possibly the utility of tests on cervical mucus samples in diagnosing endometrial cancer.

OUTLINE: This is a multicenter study. Patients are stratified by center and menopausal status. Patients are randomized to 1 of 2 arms.

* Arm I: Patients undergo insertion of the Mirena® intrauterine device containing levonorgestrel. The device is scheduled to remain in place for 4 years. Patients also undergo observation comprising an assessment of menstrual history, transvaginal scanning (TVS), and endometrial biopsy (or hysteroscopy) at baseline and then annually for 4 years.
* Arm II: Patients undergo observation comprising an assessment of menstrual history, TVS, and endometrial biopsy (or hysteroscopy) at baseline and then annually for 4 years.

Patients complete a personal health and lifestyle questionnaire, the Life Events Scale, and the Profile of Mood States (POMS) questionnaires at baseline and periodically during study.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Proven to carry a pathogenic germline mutation in a DNA mismatch repair gene causing Lynch syndrome (hereditary non-polyposis colorectal cancer) (usually MSH2, MLH1, or MSH6)
* Meets both of the following criteria:

  * Has a family history of Lynch syndrome according to the following Amsterdam or modified Amsterdam criteria:

    * Three relatives with a Lynch syndrome-related cancer (colorectal, small bowel, endometrial, ovarian, urothelial, or hepatobiliary)
    * One is a first-degree relative of the other two
    * Two generations affected
    * One relative diagnosed before age of 50
  * Personal history of colorectal cancer (i.e., a large, villous, or severely dysplastic colorectal adenoma) before the age of 40 OR history of small bowel, hepatobiliary, or urothelial cancer AND has an affected family member with an abnormal tumor immunohistochemistry staining for Lynch syndrome
* No active genital malignancy, breast carcinoma, or other estrogen dependent tumor

  * History of genital malignancy, breast carcinoma, or other estrogen dependent tumor allowed at the discretion of the investigator

PATIENT CHARACTERISTICS:

* Must have an intact uterus and not planning to undergo a prophylactic hysterectomy
* Not pregnant
* Not planning to become pregnant within the next 3 years
* No abortion resulting in infection within the past 3 months
* No pelvic inflammatory disease (PID) within the past 6 months or recurrent PID
* No clinically significant submucous myomas requiring treatment

  * Small subserous or intramural myomas, clinically assessed as insignificant allowed
* No known hypersensitivity to the constituents of the Mirena® IUS
* No unresolved abnormal cervical smear and/or current cervical dysplasia
* No trophoblastic disease with elevated hCG levels
* No liver tumor or other acute or severe liver disease
* No clinically significant condition or laboratory result that might, in the opinion of the investigator, compromise patient safety, interfere with evaluations, or prevent completion of the study
* No other active malignancy
* No history of stroke or myocardial infarction
* No history of bacterial endocarditis or severe pelvic infection after any prosthetic valve replacement or in patients with an anatomical lesion of the heart

PRIOR CONCURRENT THERAPY:

* No other concurrent use of intrauterine devices
* No concurrent therapy for cancer

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Rate of atypical endometrial hyperplasia or endometrial cancer during the active follow-up period of the study

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Hodgson, MD, Principal Investigator — St George's, University of London
Locations (20):
- United Kingdom (20):
  - Basildon University Hospital, Basildon, England
  - City Hospital - Birmingham, Birmingham, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cheltenham General Hospital, Cheltenham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead-Tyne and Wear, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Liverpool Women's Hospital, Liverpool, England
  - Guy's Hospital, London, England
  - Chelsea Westminster Hospital, London, England
  - St. Georges, University of London, London, England
  - Elizabeth Garrett Anderson Hospital, London, England
  - St. Mary's Hospital, Manchester, England
  - Royal Marsden - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - University Hospital of Wales, Cardiff, Wales